CLINICAL TRIAL: NCT05291572
Title: Comparative Study Between Three Different Methods for Stuttering Therapy in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alzahraa Momen Abdelnaeem, assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-03-02
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Stuttering, Childhood
MeSH Terms: conditions — Stuttering | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Active Comparator): will be treated by speech therapy only (fluency shaping).
  Interventions: Behavioral: speech therapy only
- Group B (Active Comparator): will be treated by speech therapy (fluency shaping) plus Hyperbaric oxygen therapy.
  Interventions: Behavioral: speech therapy only; Device: hyperbaric oxygen therapy
- Group C (Active Comparator): will be treated by speech therapy (fluency shaping) plus medical treatment (brain stimulant).
  Interventions: Behavioral: speech therapy only; Drug: medical treatment

INTERVENTIONS:
Behavioral: speech therapy only — fluency shaping technique
Device: hyperbaric oxygen therapy — chamber system using oxygen with pressure
  Arms: Group B
Drug: medical treatment — brain stimulant
  Arms: Group C

SUMMARY:
The aim of work is comparing between three different methods for treatment of stuttering in children in order to reach to the best method for treatment

ELIGIBILITY:
Inclusion Criteria:

* Children from 5 to 15 years old with IQ above 80

Exclusion Criteria:

* 1 - mental disability. 2- psychiatric problem as autism or attention deficit hyperactive disease. 3. secondary stuttering. 4. Children with sever anxiety. 5. Children with history suggested epileptic fits.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Stuttering severity instrument (SSI-3) | before therapy
  rating scale for stuttering severity

SECONDARY OUTCOMES:
Stuttering severity instrument (SSI-3) | post therapy by 3 months
  rating scale for stuttering severity